CLINICAL TRIAL: NCT05868811
Title: A Feasibility Study of Music and Play to Enhance Health and Developmental Outcomes in Infants From Low-income Families
Brief Title: Music and Child Health and Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Kansas Medical Center (Other); University of Kansas (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Kai Ling Kong, Doctoral Research Faculty, PhD, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00002451; UL1TR002366 (NIH)
Record Dates: First submitted 2023-04-20; First posted 2023-05-22 (Actual); Results first posted 2025-09-03 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Obesity, Infant; Language Development; Parent-Child Relations
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Together (Experimental)
  Interventions: Behavioral: Music Together
- Play Group (Placebo Comparator)
  Interventions: Behavioral: Play Group

INTERVENTIONS:
Behavioral: Music Together — The intervention consists of 45-minute weekly classes for 16 weeks. Each class is delivered by a trained Music Together facilitator and includes music activities such as singing, dancing, moving and playing musical instruments. At the start of the program, participants receive materials for home use that consist of a song book and online access code for song recordings used in the class.
  Arms: Music Together
Behavioral: Play Group — The play group consists of 45-minute weekly classes for 16 weeks. During each class parents are encouraged to play with their child and interact with other participants using the provided age appropriate toys. At the start of the program participants receive an age appropriate toy for use at home.
  Arms: Play Group

SUMMARY:
The goal of this clinical trial is to learn about the effects of a music enrichment program on the quality of parent child interactions, a child's motivation to eat, and a child's language environment in 9 to 24 month-old children from low-income families. The main questions it aims to answer are:

1. Does participation in a music enrichment program improve the quality of parent-child interactions?
2. Does participation in a music enrichment program reduce motivation for food
3. Does participation in a music enrichment program improve the quality of the language environment?

Participants will:

1. Be randomly assigned to participate in either 2, 8-week semesters of weekly music enrichment classes or play group sessions.
2. At the beginning, after the first 8 weeks and after the second 8 weeks, a researcher will come to the participants house and parent-child pairs will:

   1. be video recorded during 10 minutes of playtime and meal time.
   2. fill out questionnaires
   3. wear a small wearable language recorder for 16 hours
3. At the beginning, after the first 8 weeks and after the second 8 weeks, the parent and child will come to the baby lab and will:

   1. Play a computer game to test motivation for food
   2. have height and weight measurements collected

Researchers will compare the music and play groups to see if there is a difference in the quality of parent child interaction, food motivation or language environment.

ELIGIBILITY:
Inclusion Criteria:

* Family income meets criteria for the National Women, Infant, and Children (WIC) program
* Family is able and willing to commit to a 6-month program

Exclusion Criteria:

* Mother <18 years old at the time of delivery
* During pregnancy:
* Mother smoked >10 cigarettes/day
* Mother used >1 marijuana joint/day
* Mother used any other illicit drugs
* Mother drank > 3 standard drinks on a single occasion or >1 standard drink on a daily basis
* Preterm birth <37 weeks gestation
* Child with significant health issues, and/or genetic conditions (e.g., cerebral palsy, down's syndrome)
* Mother with major health concerns during pregnancy (e.g., gestational diabetes, pre-eclampsia, etc)
* Parent/child who do not speak English

Ages: 9 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kai Ling Kong, PhD, Principal Investigator — Children's Mercy
Locations (1):
- ChildrensMHC, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kong KL, Smith AR, Salley B, Hanson-Abromeit D, Engel H, Serwatka CA. A Feasibility Study of a Music Enrichment Program on Relative Reinforcing Value of Food and Home Environmental Enrichment among Families of Low Socioeconomic Status. Children (Basel). 2024 Oct 11;11(10):1229. doi: 10.3390/children11101229. PMID 39457194

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Protocol Enrollment represents the total number of dyads enrolled.
Pre-assignment Details: 4 participants dropped out after enrollment before group assignment.
Groups:
- Music Together-child: Music Together-child: The intervention consists of 45-minute weekly classes for 16 weeks. Each class is delivered by a trained Music Together facilitator and includes music activities such as singing, dancing, moving and playing musical instruments. At the start of the program, participants receive materials for home use that consist of a song book and online access code for song recordings used in the class.
- Play Group-child: Play Group-child: The play group consists of 45-minute weekly classes for 16 weeks. During each class parents are encouraged to play with their child and interact with other participants using the provided age appropriate toys. At the start of the program participants receive an age appropriate toy for use at home.
- Music Together- Parent: Music Together-parent: The intervention consists of 45-minute weekly classes for 16 weeks. Each class is delivered by a trained Music Together facilitator and includes music activities such as singing, dancing, moving and playing musical instruments. At the start of the program, participants receive materials for home use that consist of a song book and online access code for song recordings used in the class.
- Play Group- Parent: Play Group-parent: The play group consists of 45-minute weekly classes for 16 weeks. During each class parents are encouraged to play with their child and interact with other participants using the provided age appropriate toys. At the start of the program participants receive an age appropriate toy for use at home.
Period: Overall Study
Arm/Group | Music Together-child | Play Group-child | Music Together- Parent | Play Group- Parent
Started | 8 | 8 | 8 | 8
Completed | 4 | 4 | 4 | 4
Not Completed | 4 | 4 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Music Together-parent: Music Together-parent: The intervention consists of 45-minute weekly classes for 16 weeks. Each class is delivered by a trained Music Together facilitator and includes music activities such as singing, dancing, moving and playing musical instruments. At the start of the program, participants receive materials for home use that consist of a song book and online access code for song recordings used in the class.
- Play Group-parent: Play Group-parent: The play group consists of 45-minute weekly classes for 16 weeks. During each class parents are encouraged to play with their child and interact with other participants using the provided age appropriate toys. At the start of the program participants receive an age appropriate toy for use at home.
- Total: Total of all reporting groups
Arm/Group | Music Together-child | Play Group-child | Music Together-parent | Play Group-parent | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 8 | 0 | 0 | 16
  Between 18 and 65 years | 0 | 0 | 8 | 8 | 16
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.32 (0.40) | 1.43 (0.39) | 30.43 (5.02) | 33.25 (5.06) | 16.61 (2.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8 | 8 | 24
  Male | 4 | 4 | 0 | 0 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 7 | 8 | 7 | 8 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 7 | 3 | 6 | 19
  White | 3 | 0 | 4 | 1 | 8
  More than one race | 2 | 1 | 1 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 8 | 16
Relative reinforcing value of food (RRVfood) [Mean (Standard Deviation); unit: units on a scale] — RRVfood is the score for food divided by the total score (food + music). Scale range is 0-1. Lower number is the better outcome.
  The score for food is determined by a computer game to test motivation for food.
  The score for music is determined by a computer game to test motivation for music. Population: Parents were not assessed for this Baseline Measure.
  units on a scale
    number analyzed (Participants) | 8 | 8 | 0 | 0 | 16
    (all) | 0.50 (0.06) | 0.40 (0.06) |  |  | 0.45 (0.06)
Conversational turns [Mean (Standard Deviation); unit: count] — Population: Parents were not assessed for this Baseline Measure.
  count
    number analyzed (Participants) | 8 | 8 | 0 | 0 | 16
    (all) | 280.19 (69.99) | 216.07 (74.82) |  |  | 248.13 (72.41)
Use of music at home [Mean (Standard Deviation); unit: units on a scale] — Participant score is based on a questionnaire with 18 questions each with a range of 1-7. Total score range of the questionnaire is 7- 126. The higher outcome is better. Population: Parents were not assessed for this Baseline Measure.
  units on a scale
    number analyzed (Participants) | 8 | 8 | 0 | 0 | 16
    (all) | 94.87 (7.25) | 98.83 (8.26) |  |  | 96.85 (7.76)

OUTCOME MEASURES:

1. Primary Outcome: Relative Reinforcing Value of Food (RRV) Task
Description: RRVfood is a proximal measure of obesity risk. It measures how motivated one is to work to gain access to food versus non-food activity.
  RRVfood is the score for food divided by the total score (food + music). Scale range is 0-1. Lower number is the better outcome.
  The score for food is determined by a computer game to test motivation for food.
  The score for music is determined by a computer game to test motivation for music.
Time Frame: Baseline, Mid (8 weeks), Post (16 weeks)
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Music Together Baseline; Music Together Mid; Music Together Post: Music Together: The intervention consists of 45-minute weekly classes for 16 weeks. Each class is delivered by a trained Music Together facilitator and includes music activities such as singing, dancing, moving and playing musical instruments. At the start of the program, participants receive materials for home use that consist of a song book and online access code for song recordings used in the class.
- Play Group Baseline; Play Group Mid; Play Group Post: Play Group: The play group consists of 45-minute weekly classes for 16 weeks. During each class parents are encouraged to play with their child and interact with other participants using the provided age appropriate toys. At the start of the program participants receive an age appropriate toy for use at home.
Arm/Group | Music Together Baseline | Play Group Baseline | Music Together Mid | Play Group Mid | Music Together Post | Play Group Post
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
units on a scale | 0.48 (0.08) | 0.35 (0.08) | 0.5 (0.07) | 0.4 (0.07) | 0.53 (0.08) | 0.62 (0.08)

2. Primary Outcome: Use of Music at Home
Description: The Music @ Home Questionnaire was used to quantitatively assess the range of musical behaviors occurring in the home environment of families with young children.
  Participant score is based on a questionnaire with 18 questions each with a range of 1-7. Total score range of the questionnaire is 7- 126. The higher outcome is better.
Time Frame: Baseline and Post (16 weeks)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Music Together Baseline | Play Group Baseline | Music Together Post | Play Group Post
Number analyzed (Participants) | 8 | 8 | 8 | 8
units on a scale | 95 (14) | 100.5 (12.13) | 106.33 (11.33) | 98.25 (9.81)

3. Primary Outcome: Conversational Turns
Description: Back-and-forth vocalizations between a parent and child, even with pre-linguistic children, are considered a pivotal component of a high-quality early language environment because they associate with growth in specific brain regions responsible for language and cognitive development.
Time Frame: Baseline, Mid (8 weeks), Post (16 weeks)
Measure: Mean (Standard Error); unit: count
Arm/Group | Music Together Baseline | Play Group Baseline | Music Together Mid | Play Group Mid | Music Together Post | Play Group Post
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
count | 8392.67 (1625.78) | 13535.00 (1407.96) | 6116.33 (1867.00) | 13410.88 (1616.87) | 9974.50 (4227.72) | 10913.88 (3661.32)

ADVERSE EVENTS:
Time Frame: Baseline to completion of study (16 weeks).
Description: No adverse event was reported.
Arm/Group | Music Together | Play Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

LIMITATIONS AND CAVEATS:
As a pilot study, we did not power this study to detect effects on the RRVfood and home environment enrichment measures. Instead, our larger goal for this study was feasibility and acceptability. As such, our findings should be interpreted with caution and replicated in a larger sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT05868811/Prot_SAP_000.pdf